CLINICAL TRIAL: NCT02385331
Title: Molecular Mechanism of Neutrophil Necroptosis and Its Roles in RA Pathogenesis
Acronym: MMNNIRP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Principal Investigator, Hongyu Jie, Dr. Hongyu,Jie, The Third Affiliated Hospital of Southern Medical University
Other Study IDs: 201501004
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Neutrophils; necroptosis; apoptosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Neutrophils play a central role in innate immunity and are rapidly recruited to sites of infection and injury. Neutrophil apoptosis and necroptosis are essential for the inflammatory.This study is designed to investigate the cells and the molecular mechanisms of neutrophil necroptosis and apoptosis.

DETAILED DESCRIPTION:
Necrosis has recently been demonstrated to be programmatic and energy comsuming, a process termed necroptosis.

In this project, the investigators aim to investigate the mechanisms and the effects ofneutrophil necroptosis and apoptosis: 1. to investigate the cells and the molecular mechanisms that induce neutrophil necroptosis or delay apoptosis, mainly focusing on the roles of HMGB-1,TNF-α and LPS, 2. to illustrate the effects of some molecules such as TLR, TNFR, RIP1/RIP3, Caspase8, ATP and ROS in the process of sigal transduction and membrane damage during necroptosis or apoptosis , 3. to identify the similarities and differences between traditional necrosis and necroptosis in the aspects of morphologigical changes and inflammatory cytokine release, 4. to find out the effects and mechanisms of neutrophil necroptosis or apoptosis in a rheumatoid arthritis mouse model and the therapeutic effect of blocking one or several pathways in the pathogenesis of rheumatoid arthritis.

This study will not only unravel the mechanisms of neutrophil necroptosis and apoptosis, elucidate its roles and significances in inflammation and infection, but also shed new light on anti-inflammatory and anti-infection therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* age 18-65.

Exclusion Criteria:

* Don't agree with informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers，age 18-65.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-09 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The apopotosis and necroptosis of Neutrophils | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ew Sun, doctor, Study Director — Third Affiliated Hospital of Southern Medical University
Locations (1):
- Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China